CLINICAL TRIAL: NCT00839670
Title: Effects of a Modified Constraint Induced Therapy Intervention in Stroke Patients: A Multicenter, Randomized Controlled Trial.
Brief Title: Light Constraint Induced Therapy Experiment
Acronym: LICITE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: departure of the investigator coordinator into other country
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P070161
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2009-02

CONDITIONS: Stroke
Keywords: 1- Constraint induced therapy; 2- Stroke; 3- Upper limb; 4- Rehabilitation; 5- Motor training; 1- First time clinical ischemic or hemorrhagic stroke; 2- At least 10° of active wrist extension; 3- At least 10° of thumb abduction/ extension; 4- At least 10° of extension in at least 2 additional digits; 3- Adequate balance while wearing the restraint.
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Therapy (Active Comparator)
  Interventions: Other: Light constraint induced therapy
- Standard Therapy (Active Comparator)
  Interventions: Other: Standard constraint induced therapy

INTERVENTIONS:
Other: Light constraint induced therapy — 90 minutes of motor training with a physical or occupational therapist and 270 minutes of self-rehabilitation, 5 days/week/2 weeks.
  Other Names: Modified constraint induced therapy
  Arms: Modified Therapy
Other: Standard constraint induced therapy — 360 minutes of motor training with a physical or occupational therapist, 5 days/week/2 weeks
  Other Names: Constraint induced therapy
  Arms: Standard Therapy

SUMMARY:
The purpose of this trial is to compare the effect of a modified constraint induced therapy to the treatment described originally by Taub et al.. This study will determine if LICITE will lead to similar improvements than the original described method.

DETAILED DESCRIPTION:
Constraint-Induced Movement therapy or CI therapy is a rehabilitation method, that has been shown in controlled studies to produce improvements of upper limb motor function in stroke patients. However, in the original method, 6 hours of daily training are requested, which is often impossible to apply in the majority of rehabilitation unit.

The aim of this trial is to compare the effect of a modified constraint induced therapy (90 minutes of motor training with a physical or occupational therapist and 270 minutes of self-rehabilitation) to the treatment described originally by Taub et al. (360 minutes of motor training with a physical or occupational therapist).

Patients randomly received one of the two treatment and be evaluated pre- post- and 3 months after the intervention ended. The treatment will last two weeks, five days per week. The evaluations will include clinical measure of motor function and functional MRI of the brain. The brain activity will be measure just before and after the intervention with a manual motor task in order to asses brain plasticity.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age > 18 years
* First ischemic or hemorrhagic stroke between 2 and 12 months
* at least 10°of active wrist extension and at least 10° of thumb abduction/ extension, and at least 10° of extension in at least 2 additional digits.
* adequate balance while wearing the restraint

EXCLUSION CRITERIA:

* Major cognitive impairment
* Prior stroke
* Excessive fatigability
* Severe aphasia
* MAL score ≥ 2,5
* Specific exclusion criteria for fMRI ancillary study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Motor activity log scale | 10 days before inclusion, 10 days and 3 months after treatment achievement

SECONDARY OUTCOMES:
Wolf Motor Function test Stroke impact scale Functional MRI HAD scale | 10 days before inclusion, 10 days and 3 months after treatment achievement except for fMRI (no evaluation at 3 month)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SIMON, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Physique et de Réadaptation - Hôpital BICHAT, Paris, Paris Cedex 18, France